CLINICAL TRIAL: NCT05254704
Title: Validation of the French Version of the TEX-Q Questionnaire to Assess Patient's Expectations Regarding Their Surgery and Their Anesthesia.
Brief Title: Validation of the French Version of the TEX-Q Questionnaire.
Acronym: TEX-Q-F
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-A03229-32
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Expectations; Anesthesia; Surgery; Quality of Life; Patient Satisfaction; Anesthesia Awareness
Keywords: Scheduled surgery; Quality of Recovery
MeSH Terms: conditions — Patient Satisfaction; Intraoperative Awareness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group - assessment of reproductibility of TEX-Q-F: This groupe will fill in the questionnaire twice :
  * at first before the anesthesia consultation
  * then, 7 days after the consultation (without further information) This group will be composed of 100 subjects.
  We will then assess the influence of their answers on their recovery by collecting their answer of QoR-15 (quality of recovery) and EVAN-G (satisfaction) at 24 hours after the surgery.
  Interventions: Other: TEX-Q-F before scheduled surgery
- Group - assessment of the responsiveness of the questionnaire after information: This group will also fill in the questionnaire twice :
  * at first before the anesthesia consultation
  * then, 7 days after the consultation and AFTER a phone interview (about 15 minutes) with an experienced practitioner to provide appropriate information concerning the anesthesia and the postoperative rehabilitation process.
  This group will also be composed of 100 subjects.
  We will then assess the influence of their answers on their recovery by collecting their answer of QoR-15 (quality of recovery) and EVAN-G (satisfaction) at 24 hours after the surgery.
  Interventions: Other: TEX-Q-F before scheduled surgery

INTERVENTIONS:
Other: TEX-Q-F before scheduled surgery — The TEX-Q-F questionnaire (French version of the breif version of the TEX-Q) contains 15 questions to assess the patient's overall expectations concerning the surgery.
  The first 11 questions concern the patient's expectations regarding the postoperative period: pain and functional recovery. The last 4 questions focus on the patient's hopes for the outcome of the surgery. Each item is scored from 0 to 10, according to the intensity of the level of expectation.

SUMMARY:
It is now known that the level of patients' expectations about a treatment (intervention, medication) can influence their prognosis. Positive expectations impact the effectiveness of the intervention, while negative expectations may lead to adverse events.

It would therefore be useful to measure these expectations. However, there is no standardized questionnaire to report the overall level of expectation in the pre-operative phase.

A team (led by Pr Meike C Shedden-Mora) has recently developed a questionnaire that aims to assess a patient's general level of expectation regarding a therapeutic intervention, taking into account the direct benefits and the expected adverse effects. This questionnaire, the brief version of the treatment expectation questionnaire (TEX-Q) is composed of 15 items.

There's currently no French translation of the TEX-Q, nor has it been tested on a population scheduled for surgery.

In addition to expectations regarding the surgical procedure, patients seem to have various expectations regarding the impact and specific role of anesthesia. Little literature exists on specific expectations regarding the role of anesthesia.

Thus, we believe it is necessary to validate a French version of the TEX-Q questionnaire (TEX-Q-F) applied to the context of scheduled surgery, as well as to evaluate the specific expectations of anesthesia.

DETAILED DESCRIPTION:
Patients' treatment expectations are an important predictor of the impact of a therapeutic intervention (medical or psychological).

They can induce subjective and psychological changes, constituting a central mechanism of placebo and nocebo effects. Positive expectations influence the effectiveness of the intervention, whereas negative expectations may lead to adverse events. This finding also appears to be true in surgery, with a level of preoperative expectation appearing to be associated with postoperative quality of life.

The large number of existing scales measuring treatment expectancy has been identified as an important limitation to the expansion of the use of these tools. Indeed, most of them are restricted to use for a specific condition or intervention, or even focus on only one facet of expectations (either positive or negative). This observation is even more true in the field of surgery, where a recent systematic review reports that there is currently no standardised questionnaire to report the level of expectation in the preoperative phase.

A team has recently developed a questionnaire that aims to assess, in a general way, the degree of expectation of a patient regarding a therapeutic intervention, taking into account the direct benefits and undesirable effects expected through an impact that would be positive or negative. This questionnaire is composed of 35 items rated from 0 to 10 and assessing several dimensions of expectations. It was developed in English and German.

Since then, this team has developed a shorter version of the questionnaire (15 items scored from 0 to 10) to facilitate its clinical use, for which the psychometric parameters have been validated (article submitted).

So far, no French translation of this general assessment scale has been validated, nor has it been tested on a population scheduled for surgery. Similarly, until now, no evaluation of the association between the degree of preoperative expectations and the quality of post-operative recovery has been studied.

Furthermore, beyond expectations regarding the surgical procedure, patients seem to have expectations regarding the impact and the specific role of anesthesia. These expectations seem to be various and sometimes complex (not to feel nausea or pain, stay awake as much as possible, be sedated not to retain any memory of their procedure, and so on...). For example, although a Swedish team has shown that the experience of post-operative pain is correlated with the level of preoperative expectation, there is little literature on specific expectations regarding anesthesia.

Thus, it seems necessary to validate a French version of the simplified TEX-Q questionnaire (TEX-Q-F) applied to the context of scheduled surgery, as well as to evaluate the specific expectations of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years);
* Admitted for scheduled surgery in the surgical areas of orthopaedics, visceral surgery (excluding colonoscopy), neurosurgery (excluding intracranial surgery), urological, gynaecological, maxillofacial and ear, nose and throat (ENT) surgery.
* French speaking ;
* Able to answer the questionnaires, alone or with the help of a third party;
* Willing to participate in the study.
* Not suffering from a psychiatric or neurological pathology compromising cooperation with the protocol,
* Patients not already included in the study during a previous surgery,
* Date of surgery scheduled more than 7 days after the date of the anesthesia consultation,
* Non-pregnant women.

Exclusion Criteria:

* Withdrawing of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient scheduled for a surgery in the University Hospital of Angers, excepted intracranial surgery, cardiac surgery, or surgery wfor which the evaluation at 24 hours after surgery could be complicated.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Validation of the french version of the TEX-Q. | At the anesthesia consultation (One month before surgery)
  Evaluate the validity of the French version of the brief version of the TEX-Q to assess preoperative expectations before scheduled surgery

SECONDARY OUTCOMES:
Assessment of the association between expectations and the quality of postoperative recovery. | At 24 hours after surgery
  Evaluation by answering French version of quality of recovery score (QoR-15), ranged between 0 (lowest value) and 150 (highest value)
Assessment of the association between expectations and patient's satisfaction about the care provided. | At 24 hours after surgery
  Evaluation by answering EVAN-G questionnaire, composed of 26 items and 6 dimensions. . Each dimension was named according to its constitutive items: attention (5 items), privacy (4 items), information (5 items), pain (5 items), discomfort (5 items), and waiting (2 items). Items were answered using a five-point Likert scale, where 1 was much less than expected, 2 was less than expected, 3 was expected, 4 was more than expected, and 5 was much more than expected. The scores for negatively worded items were reversed so that higher scores indicated a higher level of satisfaction. the score of each dimension was obtained by computing the mean of the item scores of the dimension. All dimension scores were linearly transformed to a 0-100 scale, with 100 indicating the best possible level of satisfaction and 0 indicating the worst. The global satisfaction score was computed as the mean of the dimension scores
Minimal important difference | At the anesthesia consultation (One month before surgery)
  Estimate minimal important difference from the TEX-Q-F questionnaire in the surgery population.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alberts J, Lowe B, Glahn MA, Petrie K, Laferton J, Nestoriuc Y, Shedden-Mora M. Development of the generic, multidimensional Treatment Expectation Questionnaire (TEX-Q) through systematic literature review, expert surveys and qualitative interviews. BMJ Open. 2020 Aug 20;10(8):e036169. doi: 10.1136/bmjopen-2019-036169. PMID 32819942